CLINICAL TRIAL: NCT04000386
Title: A Study of Efficacy of Zinc Oxide Nanoparticles Coated Socks in Prevention of Unpleasant Foot Odor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: zincoxide_PK
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Zinc Oxide; Foot Dermatoses
Keywords: Pitted keratolysis; zinc oxide; Foot Odor; preventsion
MeSH Terms: conditions — Foot Dermatoses

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant) Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Single blind controlled trial between participants, drug preparing team, doctors, investigators, and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zinc oxide nanoparticles coated socks (Experimental): 62 patients with zinc oxide nanoparticles coated socks
  Interventions: Other: zinc oxide nanoparticles coated socks
- placebo (Placebo Comparator): 62 patients with placebo socks
  Interventions: Other: placebo socks

INTERVENTIONS:
Other: zinc oxide nanoparticles coated socks — zinc oxide nanoparticles coated socks were given to subjects for 2 weeks
  Arms: zinc oxide nanoparticles coated socks
Other: placebo socks — placebo socks were given to subjects for 2 weeks
  Arms: placebo

SUMMARY:
This study aimed to study the efficacy of zinc oxide nanoparticles coated socks in prevention of unpleasant foot odor

DETAILED DESCRIPTION:
Introduction Pitted keratolysis is a common skin disease, caused by various gram-positive bacteria including Corynebacterium species, Kytococcus sedentarius, Dermatophilus congolensis and Actinomyces species. These bacteria create small tunnels in the stratum corneum, causing pitted lesions at plantar areas. This condition is frequent accompanied by feet malodor and is commonly found in young male adults, especially in soldiers, miners and athletes. The reported prevalence of pitted keratolysis among naval cadets in Thailand was 38.7%. Predisposing factors related to pitted keratolysis are pedal hyperhidrosis and prolonged feet occlusion. Although this condition is generally not painful, our previous study in 2018 revealed adversely affects patients' quality of life.

Regarding treatment modalities of pitted keratolysis, various medications and life-style modification have been recommended. Previous studies revealed efficacy of topical choices, including benzoyl peroxide gel, clindamycin-benzoyl peroxide gel, glycopyrrolate cream, erythromycin gel, clindamycin solution, chlorhexidine scrub4 and mupirocin ointment. Oral antibiotics and botulinum toxin injection were also beneficial in pitted keratolysis. As to life-style modification, wearing cotton socks and opened footwear, and proper hygiene, have also been suggested.

Previous studies demonstrated efficacy of zinc oxide in broad-spectrum antibacterial properties. Thus, zinc oxide has been used in various medical and apparel industrial products. Moreover, Commander Choopong Chailark invented socks coated with zinc oxide nanoparticles and reported antibacterial property of those socks.

Objective The present study aimed to study the efficacy of zinc oxide nanoparticles coated socks in prevention of unpleasant foot odor

Material and Methods First-year naval rating cadets, who had no pedal malodor were invited to enroll in this study. Consent was informed and obtained from all participants. Participants were assessed for behavioral risk factors and level of foot odor measured by a self-assessed visual analogue scale (VAS), using questionnaires. Subjects were randomly assigned either zinc oxide nanoparticles coated socks or ordinary socks.During the study, using of other topical treatment such as topical antibiotics, antiperspirant or aluminum chloride was not allowed. Participants were advised to wear those socks every day and regularly washed thier socks. All were able to regularly participate in physical military training during the study. Two weeks after the study clinical examinations by dermatologists and the cadets' self-assessment questionnaires, including feet odor by using VAS, treatment satisfaction and adverse effects, were used to evaluate the effectiveness. Pitted lesions improvement at plantar areas, evaluated by dermatologists, was divided into no improvement, slight improvement (decrease of pitted lesions at feet for 1 level) and much improvement (decrease of pitted lesions at feet for at least 2 level). Data were analyzed using Predictive Analytics SoftWare Statistics version 18 (SPSS, Inc., Chicago, Illinois, USA).

Duration of study: 4 months

Study design: Randomized control trial

ELIGIBILITY:
Inclusion Criteria:

* First-year naval rating cadets, who had no pedal malodor

Exclusion Criteria:

* The cadets who previously received any topical treatment including topical antibiotic, antiperspirant or aluminum chloride within 6 months prior to the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Effectiveness of zinc oxide nanoparticles coated socks in prevention of unpleasant foot odor | 2 weeks
  Effectiveness was evaluated by the number of patients who had no or minimal foot odor after prevention

SECONDARY OUTCOMES:
Effectiveness of zinc oxide nanoparticles coated socks in prevention of fungal feet infection | 2 weeks
  Effectiveness was evaluated by the number of patients who had no fungal feet infection after prevention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] de Almeida HL Jr, Siqueira RN, Meireles Rda S, Rampon G, de Castro LA, Silva RM. Pitted keratolysis. An Bras Dermatol. 2016 Jan-Feb;91(1):106-8. doi: 10.1590/abd1806-4841.20164096. PMID 26982791
- [Result] Makhecha M, Dass S, Singh T, Gandhi R, Yadav T, Rathod D. Pitted keratolysis - a study of various clinical manifestations. Int J Dermatol. 2017 Nov;56(11):1154-1160. doi: 10.1111/ijd.13744. Epub 2017 Sep 18. PMID 28924971
- [Result] van der Snoek EM, Ekkelenkamp MB, Suykerbuyk JC. Pitted keratolysis; physicians' treatment and their perceptions in Dutch army personnel. J Eur Acad Dermatol Venereol. 2013 Sep;27(9):1120-6. doi: 10.1111/j.1468-3083.2012.04674.x. Epub 2012 Aug 7. PMID 22882561
- [Result] Leeyaphan C, Bunyaratavej S, Taychakhoonavudh S, Kulthanachairojana N, Pattanaprichakul P, Chanyachailert P, Ongsri P, Arunkajohnsak S, Limphoka P, Kulthanan K. Cost-effectiveness analysis and safety of erythromycin 4% gel and 4% chlorhexidine scrub for pitted keratolysis treatment. J Dermatolog Treat. 2019 Sep;30(6):627-629. doi: 10.1080/09546634.2018.1543846. Epub 2018 Dec 11. PMID 30415588
- [Result] Vlahovic TC, Dunn SP, Kemp K. The use of a clindamycin 1%-benzoyl peroxide 5% topical gel in the treatment of pitted keratolysis: a novel therapy. Adv Skin Wound Care. 2009 Dec;22(12):564-6. doi: 10.1097/01.ASW.0000363468.18117.fe. No abstract available. PMID 19935134
- [Result] Bunyaratavej S, Leeyaphan C, Chanyachailert P, Pattanaprichakul P, Ongsri P, Kulthanan K. Clinical manifestations, risk factors and quality of life in patients with pitted keratolysis: a cross-sectional study in cadets. Br J Dermatol. 2018 Nov;179(5):1220-1221. doi: 10.1111/bjd.16923. Epub 2018 Sep 14. No abstract available. PMID 29951993
- [Result] Burkhart CG. Pitted keratolysis: a new form of treatment. Arch Dermatol. 1980 Oct;116(10):1104. No abstract available. PMID 7425659
- [Result] Balic A, Bukvic Mokos Z, Marinovic B, Ledic Drvar D. Tatami Mats: A Source of Pitted Keratolysis in a Martial Arts Athlete? Acta Dermatovenerol Croat. 2018 Apr;26(1):68-70. PMID 29782305
- [Result] Kontochristopoulos G, Sidiropoulou P, Tzanetakou V, Markantoni V, Platsidaki E, Agiasofitou E, Rigopoulos D, Gregoriou S. Managing pitted keratolysis: consider topical glycopyrrolate. Clin Exp Dermatol. 2019 Aug;44(6):713-714. doi: 10.1111/ced.13851. Epub 2018 Dec 4. No abstract available. PMID 30515854
- [Result] Pranteda G, Carlesimo M, Pranteda G, Abruzzese C, Grimaldi M, De Micco S, Muscianese M, Bottoni U. Pitted keratolysis, erythromycin, and hyperhidrosis. Dermatol Ther. 2014 Mar-Apr;27(2):101-4. doi: 10.1111/dth.12064. Epub 2013 May 24. PMID 24703267
- [Result] Greywal T, Cohen PR. Pitted keratolysis: successful management with mupirocin 2% ointment monotherapy. Dermatol Online J. 2015 Aug 15;21(8):13030/qt6155v9wk. PMID 26437161
- [Result] Vazquez-Lopez F, Perez-Oliva N. Mupirocine ointment for symptomatic pitted keratolysis. Infection. 1996 Jan-Feb;24(1):55. doi: 10.1007/BF01780656. No abstract available. PMID 8852468
- [Result] Tamura BM, Cuce LC, Souza RL, Levites J. Plantar hyperhidrosis and pitted keratolysis treated with botulinum toxin injection. Dermatol Surg. 2004 Dec;30(12 Pt 2):1510-4. doi: 10.1111/j.1524-4725.2004.30553.x. PMID 15606827
- [Result] Fiedot-Tobola M, Ciesielska M, Maliszewska I, Rac-Rumijowska O, Suchorska-Wozniak P, Teterycz H, Bryjak M. Deposition of Zinc Oxide on Different Polymer Textiles and Their Antibacterial Properties. Materials (Basel). 2018 Apr 30;11(5):707. doi: 10.3390/ma11050707. PMID 29710873
- [Result] Raghunath A, Perumal E. Metal oxide nanoparticles as antimicrobial agents: a promise for the future. Int J Antimicrob Agents. 2017 Feb;49(2):137-152. doi: 10.1016/j.ijantimicag.2016.11.011. Epub 2017 Jan 3. PMID 28089172
- [Result] Dizaj SM, Lotfipour F, Barzegar-Jalali M, Zarrintan MH, Adibkia K. Antimicrobial activity of the metals and metal oxide nanoparticles. Mater Sci Eng C Mater Biol Appl. 2014 Nov;44:278-84. doi: 10.1016/j.msec.2014.08.031. Epub 2014 Aug 16. PMID 25280707